CLINICAL TRIAL: NCT02519413
Title: A Retrospective, Multi-Center, Observational Study to Assess the Effect of Tecfidera® Delayed-Release Capsules on Lymphocyte Subsets in Subjects With Relapsing Forms of Multiple Sclerosis (REALIZE)
Brief Title: Tecfidera Lymphocyte Chart Review
Acronym: REALIZE
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS419
Record Dates: First submitted 2015-07-16; First posted 2015-08-10 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis
Keywords: lymphocyte; serious infections; opportunistic infections; Relapsing Forms
MeSH Terms: conditions — Multiple Sclerosis; Opportunistic Infections | interventions — Dimethyl Fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dimethyl fumarate — delayed release capsules
  Other Names: DMF; Tecfidera; BG00012

SUMMARY:
The primary objective of the study is to retrospectively investigate changes in lymphocyte counts and lymphocyte subtypes, with a focus on CD4+ and CD8+ T cells, in participants on Tecfidera therapy for at least 6 months. The secondary objective is to investigate changes in lymphocyte subtypes other than CD4+ and CD8+ T cells.

ELIGIBILITY:
Key Inclusion Criteria:

* Initiated Tecfidera treatment for the first time on or after 27 March 2013 and received at least 6 months of continuous treatment with Tecfidera
* Clinical diagnosis of a relapsing form of MS
* A baseline measurement for ALC and absolute CD4+ or CD8+ count within 6 months prior to Tecfidera initiation
* At least 1 measurement for ALC and absolute CD4+ or CD8+ count while on Tecfidera therapy for at least 6 months

Key Exclusion Criteria:

* Clinical diagnosis of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) prior to Tecfidera initiation
* Participation in DEFINE 109MS301 (NCT00420212) or CONFIRM 109MS302 (NCT00451451)

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in patients with relapsing forms of multiple sclerosis (MS) who initiated Tecfidera treatment for the first time (treatment naïve) under routine clinical care. For inclusion in the study, patients' charts must have a baseline measurement for absolute lymphocyte count (ALC) and absolute CD4+ or CD8+ count within 6 months prior to Tecfidera initiation, and at least 1 measurement for ALC and absolute CD4+ or CD8+ count while on Tecfidera treatment for at least 6 months. For patients who discontinue Tecfidera, data will be collected for up to 6 months following Tecfidera discontinuation.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Estimated absolute lymphocyte count (ALC) change from baseline following Tecfidera initiation | 6 and 12 months
Estimated CD4+ count change from baseline following Tecfidera initiation | 6 and 12 months
Estimated CD8+ count change from baseline following Tecfidera initiation | 6 and 12 months

SECONDARY OUTCOMES:
Raw absolute counts for leukocyte, lymphocyte, CD4+/CD8+ ratio following Tecfidera initiation | 6 and 12 months
Raw absolute counts for additional lymphocyte subsets (other than CD4+ and CD8+) | 6 and 12 months
Change from baseline for leukocyte, lymphocyte, CD4+/CD8+ ratio following Tecfidera initiation | 6 and 12 months
Change from baseline for additional lymphocyte subsets (other than CD4+and CD8+) following Tecfidera initiation | 6 and 12 months
Percentage change from baseline for leukocyte, lymphocyte, CD4+/CD8+ ratio following Tecfidera initiation | 6 and 12 months
Percentage change from baseline for additional lymphocyte subsets (other than CD4+and CD8+) following Tecfidera initiation | 6 and 12 months
Time to pre-determined lymphocyte counts following Tecfidera initiation | Up to 12 months
Potential predictors of low lymphocyte counts following Tecfidera initiation | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (9):
- United States (9):
  - Research site, Homewood, Alabama
  - Research Site, Newport Beach, California
  - Research Site, Atlanta, Georgia
  - Research Site, Buffalo, New York
  - Research Site, Patchogue, New York
  - Research Site, Huntersville, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin